CLINICAL TRIAL: NCT02945514
Title: Validation of the Measurement and Prediction of the Postprandial Glycemic Response to Food and Providing Personally Tailored Dietary Recommendations
Brief Title: Providing Personally Tailored Dietary Suggestions Using Individual Microbiome and Glycemic Index Response.
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: DayTwo (Industry)
Responsible Party: Principal Investigator, Heidi Nelson, M.D., Mayo Clinic
Other Study IDs: 16-005208
Record Dates: First submitted 2016-10-24; First posted 2016-10-26 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Healthy Volunteers
Keywords: Healthy; Diet; Microbiome; Personalized; Custom

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood and Stool
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: DayTwo machine learning algorithm — Personally tailored nutrition insights based on DayTwo machine learning algorithm when combining facets of your postprandial glycemic response to food consumed during collection week and your individual gut microbiome composition

SUMMARY:
Provide personally tailored dietary suggestions to participants based on the Personalized Prediction Engine (patent pending) owned by DayTwo.

DETAILED DESCRIPTION:
* Answer personal questions including such things as health information, eating habits and preferences, activity level and intensity.
* Submit a first stool sample via a self-addressed, postage-paid kit that is mailed to you.
* Attend one of the 2 hour connection meetings based on available dates.
* The study team will collect vitals: measurements of height, weight, blood pressure, pulse, waist and hip circumference.
* You will have a Blood collection for study (approximately 35 ml of blood/5 tubes)
* You will be provided a FitBit wrist band that you will wear
* You will be provided a manual blood glucose monitor you will use for pricking finger and measuring blood sugar level at least 4 times per day.
* You will have a continuous blood glucose sensor and monitor inserted by study staff.
* You will use DayTwo's mobile application where you will input food eaten, activity, measurements, medications, and sleep.
* You will be given a second stool kit and instructions for collection.
* You will be asked to eat 4 breakfasts consisting of either bagels and cream cheese or cereal. These foods will be provided for you. Other than these four breakfasts, we would like you to follow your normal eating habits during the collection week.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Comprehension of the study objectives and requirements
* Ability to download the DayTwo proprietary mobile application
* Ability to access the DayTwo website for registration and nutrition report

Exclusion Criteria:

* Under 18 years of age
* Pre-diagnosed type I or type II diabetes mellitus
* Pregnancy
* Use of antibiotics or fertility treatments within 3 months prior to participation
* Bariatric weight loss surgery
* Chronic Anemia (hemoglobin of 10g per deciliter or less
* Chronic gastrointestinal disorder (IBD, Celiac, etc.)
* Active cancer or chemotherapy or radiation within 2 years prior to participation
* Condition not allowing to follow the dietary recommendation during the study
* 4 or more alcoholic drinks per day on a regular basis or use of recreational drugs
* Chronic medical condition, treatment, or medication that may affect glucose metabolism (HIV diagnosis, use of steroids or immunosuppressive drugs, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men and women above 18 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 327 (Actual)
Dates: Start 2016-09; Primary Completion 2018-02-27 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Postprandial blood sugar level | Baseline through 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Nelson, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zeevi D, Korem T, Zmora N, Israeli D, Rothschild D, Weinberger A, Ben-Yacov O, Lador D, Avnit-Sagi T, Lotan-Pompan M, Suez J, Mahdi JA, Matot E, Malka G, Kosower N, Rein M, Zilberman-Schapira G, Dohnalova L, Pevsner-Fischer M, Bikovsky R, Halpern Z, Elinav E, Segal E. Personalized Nutrition by Prediction of Glycemic Responses. Cell. 2015 Nov 19;163(5):1079-1094. doi: 10.1016/j.cell.2015.11.001. PMID 26590418
- [Derived] Mendes-Soares H, Raveh-Sadka T, Azulay S, Ben-Shlomo Y, Cohen Y, Ofek T, Stevens J, Bachrach D, Kashyap P, Segal L, Nelson H. Model of personalized postprandial glycemic response to food developed for an Israeli cohort predicts responses in Midwestern American individuals. Am J Clin Nutr. 2019 Jul 1;110(1):63-75. doi: 10.1093/ajcn/nqz028. PMID 31095300